CLINICAL TRIAL: NCT06802835
Title: EGFR Antibody Combined With Programmed Death-1 Inhibitor and Chemotherapy in Recurrent/Metastatic Nasopharyngeal Carcinoma: A Prospective, Multi-center, Phase I/II Clinical Trial
Brief Title: EGFR Antibody Combined With PD-1 Inhibitor and Chemotherapy in R/M Nasopharyngeal Carcinoma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Zhao Chong, Prof., Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EGFR+PD-1+Chemo for r/mNPC
Record Dates: First submitted 2025-01-25; First posted 2025-01-31 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Nasopharyngeal Cancinoma (NPC); Recurrent Nasopharynx Carcinoma; Metastatic Nasopharyngeal Carcinoma
Keywords: EGFR antibody; PD-1 antibody; chemotherapy
MeSH Terms: conditions — Nasopharyngeal Neoplasms; Nasopharyngeal Carcinoma | interventions — spartalizumab; Gemcitabine; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- EGFR+PD-1+Chemo (Experimental)
  Interventions: Drug: EGFR Antibody; Drug: PD-1 antibody; Drug: Gemcitabine, Cisplatin; Radiation: IMRT

INTERVENTIONS:
Drug: EGFR Antibody — 6 cycles for combined therapy. Maintenance for 1 year.
Drug: PD-1 antibody — 6 cycles for combined therapy. Maintenance for 1 year.
Drug: Gemcitabine, Cisplatin — 6 cycles for combined therapy.
Radiation: IMRT — IMRT for primary lesion

SUMMARY:
This is a prospective, single-arm, phase II clinical trial. The purpose of this study is to evaluate the efficacy and adverse effect of EGFR antibody combined with programmed death 1 (PD-1) antibody and chemotherapy in recurrent/metastatic nasopharyngeal carcinoma patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with nasopharyngeal carcinoma who have recurred/metastasized after initial treatment or radical treatment;
* Age 18-75, male or female;
* Pathological diagnosis of nasopharyngeal carcinoma;
* ECOG score 0-1;
* Have not previously received any anti-tumor therapy such as radiotherapy, chemotherapy, immunotherapy or biotherapy for recurrence/metastasis;
* No contraindications of chemotherapy, immunotherapy and targeted therapy;
* At least 1 measurable lesion that meets RECIST 1.1 criteria;
* Blood routine examination standards should meet: WBC≥3.0×109/L, ANC≥1.5×109/L, PLT≥100×109/L, HGB≥90g/L (no blood transfusion and blood products within 14 days, no G-CSF and other hematopoietic stimulating factors are used to correct);
* Biochemical tests should meet the following criteria: TBIL≤2.0×ULN, ALT, AST≤2.5×ULN, BUN and CRE≤1.5×ULN or endogenous creatinine clearance ≥60ml/min (Cockcroft-Gault formula);
* Good coagulation function: defined as International standardized ratio (INR) or prothrombin time (PT) ≤1.5 times ULN; If the subject is receiving anticoagulant therapy, as long as PT is within the intended range of anticoagulant drug use;
* The myocardial enzyme spectra were in the normal range;
* Women of childbearing age must already be using reliable contraception or have had a pregnancy test (serum or urine) within 7 days of enrollment with a negative result and be willing to use an effective method of contraception during the trial and for 3 months after the last anti-PD-1 antibody administration. For male subjects whose partners are women of reproductive age, effective contraception should be used during the trial and within 3 months after the last anti-PD-1 antibody administration;
* The subjects voluntarily joined the study, signed informed consent, had good compliance, and cooperated with follow-up;

Exclusion Criteria:

* Patients with recurrence who can be treated with local resection or radiotherapy;
* Known to be allergic to the investigational drug or any excipients thereof, or has had a severe allergic reaction to other monoclonal antibodies;
* Patients have symptoms of central nervous system metastasis such as brain edema and need hormonal intervention;
* Had an active infection or unexplained fever >38.5℃ during screening or prior to the first dose (the investigator determined that the subject's fever due to the tumor could be enrolled);
* Have any active autoimmune disease or history of autoimmune disease (e.g., interstitial pneumonia, uveitis, enteritis, hepatitis, hypophysitis, vasculitis, myocarditis, nephritis, hyperthyroidism, hypothyroidism [may be included after normal hormone replacement therapy]); Patients with vitiligo or complete remission of asthma in childhood without any intervention as adults could be included, but patients with asthma requiring medical intervention with bronchodilators could not be included;
* Have congenital or acquired immunodeficiency (such as HIV), active hepatitis B (HBV-DNA≥103 copy number /ml), or hepatitis C (hepatitis C antibody positive and HCR-RNA above the lower detection limit of analytical methods);
* Previous or co-existing uncured malignancies, except cured basal cell carcinoma of the skin, carcinoma in situ of the cervix and superficial bladder cancer;
* Uncontrolled cardiovascular disease: Grade II or higher myocardial ischemia or myocardial infarction, poorly controlled arrhythmias (including QTc interval ≥470 ms); Patients with grade III-IV cardiac insufficiency according to NYHA standards, or left ventricular ejection fraction (LVEF) <50% indicated by cardiac color ultrasound; Myocardial infarction within 1 year;
* If the subject has undergone major surgery, the toxic effects and/or complications of the surgical intervention must be fully recovered before treatment is initiated;
* Within 4 weeks prior to the first use of the investigational drug (participants in the follow-up period are counted as the last use of the investigational drug or device) or are currently participating in another clinical study;
* Live vaccine received within 4 weeks prior to the first administration of the investigational drug is allowed to receive inactivated virus vaccine for seasonal influenza by injection, but not live attenuated influenza vaccine for nasal administration;
* Pregnant or lactating women;
* In the investigator's judgment, the subjects had other factors that might have led to their forced discontinuation of the study, such as other serious medical conditions (including mental illness) requiring concomitant treatment, serious abnormalities in laboratory test values, or family or social factors that might have affected the safety of the subjects or the circumstances of the trial data collection.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2027-02-20 (Estimated); Study Completion 2029-02-20 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | 1 year
  From the date of recruiting to the first occurrence of disease progression as determined according to RECIST v1.1 or death from any cause, whichever occurs first.

SECONDARY OUTCOMES:
Adverse events | Up to 16 months
  All adverse event or serious adverse event that occurred during the study period according to CTCAE v 5.0.
Overall survival (OS) | 1 year
  From the date of recruiting to the date of death from any cause.
Objective response rate (ORR) | 1 year
  The percentage of patients with CR and PR assessed according to RECIST v1.1.
Disease control rate (DCR) | 1 year
  The proportion of patients who have achieved complete response, partial response and stable disease according to RECIST v1.1.
Quality of life (QoL) | 1 year
  Assessed by EQ-5D-5L questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No